CLINICAL TRIAL: NCT04519658
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter, Parallel-Group, Dose-Ranging Study to Evaluate the Efficacy and Safety of Multiple Dose Strengths of CIN-107 as Compared to Placebo After 12 Weeks of Treatment in Patients With Treatment-Resistant Hypertension (rHTN)
Brief Title: A Study of CIN-107 in Adults With Treatment-Resistant Hypertension (rHTN)
Acronym: BrigHTN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CinCor Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIN-107-121
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Resistant Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CIN-107 0.5mg (Experimental): Subjects received CIN-107 0.5 mg tablets, administered orally once daily for 12 weeks. Subjects continued taking stable anti-hypertensive regimen throughout the study.
  Interventions: Drug: CIN-107
- CIN-107 1mg (Experimental): Subjects received CIN-107 1 mg tablets, administered orally once daily for 12 weeks. Subjects continued taking stable anti-hypertensive regimen throughout the study.
  Interventions: Drug: CIN-107
- CIN-107 2mg (Experimental): Subjects received CIN-107 2 mg tablets, administered orally once daily for 12 weeks. Subjects continued taking stable anti-hypertensive regimen throughout the study.
  Interventions: Drug: CIN-107
- Placebo (Placebo Comparator): Subjects received placebo tablets, administered orally once daily for 12 weeks. Subjects continued taking stable anti-hypertensive regimen throughout the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CIN-107 — CIN-107 tablets by mouth once daily
  Other Names: baxdrostat
  Arms: CIN-107 0.5mg; CIN-107 1mg; CIN-107 2mg
Drug: Placebo — placebo tablets by mouth once daily
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, dose-ranging Phase 2 study to evaluate the efficacy and safety of CIN-107 as compared to placebo after 12 weeks of treatment in patients with treatment-resistant hypertension (rHTN).

ELIGIBILITY:
Inclusion Criteria:

* Is on a stable regimen of ≥ 3 antihypertensive agents (one of which is a diuretic) for at least 4 weeks prior to randomization;
* Be at least 70% compliant to their anti-hypertensive medication regimen;
* Has a seated BP ≥ 130/80 mmHg;
* Agrees to comply with the contraception and reproduction restrictions of the study; and
* Able to understand and willing to comply with all study visits, procedures, restrictions, and provide written informed consent according to institutional and regulatory guidelines.

Exclusion Criteria:

* Has a seated SBP ≥ 180 mmHg or DBP ≥ 110 mmHg;
* Has a body mass index (BMI) > 40 kg/m2;
* Has an upper arm circumference < 7 or > 17 inches;
* Has been on night shifts at any time during the 4 weeks before Screening;
* Is using a beta blocker for any primary indication other than systemic hypertension (eg, migraine headache);
* Is not willing or not able to discontinue an MRA or a potassium sparing diuretic as part of an existing antihypertensive regimen;
* Is not willing or not able to discontinue taking a potassium supplement;
* Has documented estimated glomerular filtration rate (eGFR) < 45 mL/min/1.73m2
* Has known and documented New York Heart Association stage III or IV chronic heart failure
* Has had a stroke, transient ischemic attack, hypertensive encephalopathy, acute coronary syndrome, or hospitalization for heart failure within 6 months before Screening;
* Has known current severe left ventricular outflow obstruction, such as obstructive hypertrophic cardiomyopathy and/or severe aortic valvular disease diagnosed from a prior echocardiogram;
* Major cardiac surgery (eg, CABG, valve replacement), peripheral arterial bypass surgery, or PCI within 6 months before Screening;
* Has chronic permanent atrial fibrillation;
* Has uncontrolled diabetes with glycosylated hemoglobin > 9.5% at Screening;
* Has planned dialysis or kidney transplant during the course of this study;
* Potassium < 3.5 mEq/L;
* Potassium > 5.0 mEq/L;
* Is positive for HIV antibody, hepatitis C virus RNA, or hepatitis B surface antigen;
* Has typical consumption of ≥14 alcoholic drinks weekly.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (80):
- United States (80):
  - CinCor Site 16, Birmingham, Alabama
  - CinCor Site 38, Birmingham, Alabama
  - CinCor Site 61, Saraland, Alabama
  - CinCor Site 90, Tucson, Arizona
  - CinCor Site 82, Anaheim, California
  - CinCor Site 91, Granada Hills, California
  - CinCor Site 25, Lincoln, California
  - CinCor Site 73, Los Angeles, California
  - CinCor Site 36, Los Angeles, California
  - CinCor Site 34, Lynwood, California
  - CinCor Site 14, San Dimas, California
  - CinCor Site 28, Santa Ana, California
  - CinCor Site 19, Spring Valley, California
  - CinCor Site 32, Tustin, California
  - CinCor Site 44, West Hills, California
  - CinCor Site 66, Whittier, California
  - CinCor Site 56, Stamford, Connecticut
  - CinCor Site 30, Clearwater, Florida
  - CinCor Site 13, Fort Myers, Florida
  - CinCor Site 74, Hialeah, Florida
  - CinCor Site 22, Homestead, Florida
  - CinCor Site 20, Jacksonville, Florida
  - CinCor Site 1, Jupiter, Florida
  - CinCor Site 84, Lake Worth, Florida
  - CinCor Site 70, Miami, Florida
  - CinCor Site 89, Miami, Florida
  - CinCor Site 94, Miami, Florida
  - CinCor Site 5, Port Orange, Florida
  - CinCor Site 9, St. Petersburg, Florida
  - CinCor Site 23, Tampa, Florida
  - CinCor Site 88, Winter Haven, Florida
  - CinCor Site 71, Suwanee, Georgia
  - CinCor Site 11, Meridian, Idaho
  - CinCor Site 15, Addison, Illinois
  - CinCor Site 81, Arlington Heights, Illinois
  - CinCor Site 49, Chicago, Illinois
  - CinCor Site 35, Morton, Illinois
  - CinCor Site 58, Evansville, Indiana
  - CinCor Site 54, West Des Moines, Iowa
  - CinCor Site 29, Lexington, Kentucky
  - CinCor Site 24, Lexington, Kentucky
  - CinCor Site 69, New Orleans, Louisiana
  - CinCor Site 64, Shreveport, Louisiana
  - CinCor Site 75, Baltimore, Maryland
  - CinCor Site 65, Elkridge, Maryland
  - CinCor Site 52, Roseville, Michigan
  - CinCor Site 21, Troy, Michigan
  - CinCor Site 92, Hattiesburg, Mississippi
  - CinCor Site 50, Olive Branch, Mississippi
  - CinCor Site 45, Butte, Montana
  - CinCor Site 47, Las Vegas, Nevada
  - CinCor Site 31, Albuquerque, New Mexico
  - CinCor Site 55, Johnson City, New York
  - CinCor Site 4, The Bronx, New York
  - CinCor Site 59, Cincinnati, Ohio
  - CinCor Site 6, Cincinnati, Ohio
  - CinCor Site 7, Cincinnati, Ohio
  - CinCor Site 86, Dayton, Ohio
  - CinCor Site 43, Beaver, Pennsylvania
  - CinCor Site 39, Myrtle Beach, South Carolina
  - CinCor Site 97, Jackson, Tennessee
  - CinCor Site 42, Knoxville, Tennessee
  - CinCor Site 27, Austin, Texas
  - CinCor Site 80, Carrollton, Texas
  - CinCor Site 79, Dallas, Texas
  - CinCor Site 87, Friendswood, Texas
  - CinCor Site 2, Houston, Texas
  - CinCor Site 72, Houston, Texas
  - CinCor Site 46, Hurst, Texas
  - CinCor Site 93, Kerville, Texas
  - CinCor Site 37, McAllen, Texas
  - CinCor Site 85, Sugar Land, Texas
  - CinCor Site 48, Draper, Utah
  - CinCor Site 3, Salt Lake City, Utah
  - CinCor Site 77, Alexandria, Virginia
  - CinCor Site 8, Burke, Virginia
  - CinCor Site 33, Manassas, Virginia
  - CinCor Site 76, Norfolk, Virginia
  - CinCor Site 41, Olympia, Washington
  - CinCor Site 51, Kenosha, Wisconsin

REFERENCES:
- [Background] Freeman MW, Halvorsen YD, Marshall W, Pater M, Isaacsohn J, Pearce C, Murphy B, Alp N, Srivastava A, Bhatt DL, Brown MJ; BrigHTN Investigators. Phase 2 Trial of Baxdrostat for Treatment-Resistant Hypertension. N Engl J Med. 2023 Feb 2;388(5):395-405. doi: 10.1056/NEJMoa2213169. Epub 2022 Nov 7. PMID 36342143

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was a 2-week Single Blind Run-In (SB-RI) period with administration of placebo before inclusion in the double-blind, randomized part of the study. 360 patients entered SB-RI and 85 patients withdrew early from SB-RI. 275 patients were randomized to 1 of the 4 treatment groups.
Groups:
- CIN-107 Dose 1 (0.5mg); CIN-107 Dose 2 (1mg); CIN-107 Dose 3 (2mg): CIN-107: CIN-107 tablets by mouth once daily
Period: Overall Study
Arm/Group | CIN-107 Dose 1 (0.5mg) | CIN-107 Dose 2 (1mg) | CIN-107 Dose 3 (2mg) | Placebo
Started | 69 | 70 | 67 | 69
Completed | 65 | 60 | 56 | 67
Not Completed | 4 | 10 | 11 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CIN-107 Dose 1 (0.5mg) | CIN-107 Dose 2 (1mg) | CIN-107 Dose 3 (2mg) | Placebo | Total
Number analyzed (Participants) | 69 | 70 | 67 | 69 | 275
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 39 | 41 | 32 | 151
  >=65 years | 30 | 31 | 26 | 37 | 124
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.5 (10.28) | 62.7 (10.14) | 61.2 (10.77) | 63.8 (10.78) | 62.3 (10.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 33 | 29 | 27 | 122
  Male | 36 | 37 | 38 | 42 | 153
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 1 | 2 | 1 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 22 | 20 | 19 | 16 | 77
  White | 45 | 48 | 47 | 51 | 191
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 69 | 70 | 67 | 69 | 275
Seated SBP [Mean (Standard Deviation); unit: mmHg] | 147.6 (12.49) | 147.7 (13.05) | 147.3 (11.82) | 148.9 (12.38) | 147.9 (12.40)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Seated Systolic BP (SBP)
Time Frame: 12 weeks
Population: Only patients with non-missing baseline and the specified visit were included.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- mITT Population 0.5mg; mITT Population 1mg; mITT Population 2mg; mITT Population Placebo: The mITT Population included all patients in the ITT Population who received at least 1 dose of any study drug and had a baseline value for the SBP assessment.
Arm/Group | mITT Population 0.5mg | mITT Population 1mg | mITT Population 2mg | mITT Population Placebo
Number analyzed (Participants) | 65 | 60 | 54 | 67
mmHg | -12.4 (15.63) | -17.3 (18.10) | -19.2 (15.84) | -9.8 (13.71)

2. Secondary Outcome: Change From Baseline in Mean Seated Diastolic BP (DBP)
Time Frame: 12 weeks
Population: Only patients with non-missing baseline and the specified visit were included.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | mITT Population 0.5mg | mITT Population 1mg | mITT Population 2mg | mITT Population Placebo
Number analyzed (Participants) | 65 | 60 | 54 | 67
mmHg | -9.1 (9.04) | -11.7 (9.88) | -14.0 (12.42) | -9.3 (9.6)

3. Secondary Outcome: The Percentage of Patients Achieving a Seated BP Response <130/80 mmHg
Time Frame: 12 weeks
Population: The modified ITT (mITT) Population included all patients in the ITT Population who received at least 1 dose of any study drug and had a baseline value for the SBP assessment. Any efficacy measurement obtained after a patient received a restricted BP altering therapy, outside of the current study design, was removed from the mITT analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | mITT Population 0.5mg | mITT Population 1mg | mITT Population 2mg | mITT Population Placebo
Number analyzed (Participants) | 69 | 69 | 67 | 69
Participants | 21 | 28 | 26 | 21

ADVERSE EVENTS:
Time Frame: From the time of informed consent to the end of the Follow-up Period, up to 24 weeks.
Description: One patient who was randomized to the 1 mg CIN-107 treatment group withdrew from the study prior to treatment with the study drug due to the physician's decision.
Groups:
- Safety Population 0.5mg; Safety Population 1mg; Safety Population 2mg; Safety Population Placebo: The Safety Population included all patients who received at least 1 dose of any randomized study drug.
Arm/Group | Safety Population 0.5mg | Safety Population 1mg | Safety Population 2mg | Safety Population Placebo
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/69 | 0/67 | 0/69
Serious Adverse Events (participants affected / at risk) | 0/69 | 2/69 | 6/67 | 2/69
Other Adverse Events (participants affected / at risk) | 6/69 | 16/69 | 8/67 | 10/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population 0.5mg (N=69) | Safety Population 1mg (N=69) | Safety Population 2mg (N=67) | Safety Population Placebo (N=69)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Safety Population 0.5mg (N=69) | Safety Population 1mg (N=69) | Safety Population 2mg (N=67) | Safety Population Placebo (N=69)
Urinary tract infection (Infections and infestations) | 3 | 7 | 6 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 5 | 2 | 1
Fatigue (General disorders) | 0 | 4 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 4
Headache (Nervous system disorders) | 1 | 5 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less or equal to 60 days from the time submitted to the sponsor for review. The sponsor can require changes to the communication and can extend the embargo for up to 90 days.

DOCUMENTS (2):
  • Study Protocol (2021-12-07): https://cdn.clinicaltrials.gov/large-docs/58/NCT04519658/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-12): https://cdn.clinicaltrials.gov/large-docs/58/NCT04519658/SAP_001.pdf